CLINICAL TRIAL: NCT03503435
Title: The Effect of Art Therapy on Psychological and Physiological Health in Total Laryngectomy Patients
Brief Title: The Effect of Art Therapy on Total Laryngectomy Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 we are not able to recruit in the foreseeable future
Sponsor: University of Haifa (Other)
Collaborators: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Johanna Czamanski-Cohen, Researcher, University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: TL-Art
Record Dates: First submitted 2018-04-11; First posted 2018-04-19 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Quality of Life; Depressive Symptoms
Keywords: Art Therapy; Total Laryngectomy
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: This is a pre and post design quasi-experimental study looking at changes before and after a supportive care art therapy intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Art therapy intervention (Other): Participants will then take part in six-weeks of group art therapy with a goal of increasing self-awareness and expression. During the intervention sessions, participants will have access to a wide range of materials conventionally used in art therapy excluding materials that may be abrasive or powdery and unsuitable around people wearing a stoma.
  Interventions: Behavioral: Group art therapy

INTERVENTIONS:
Behavioral: Group art therapy — Participants will undergo 6 weeks of group art therapy in which they will learn tools to cope with a variety of cognitive, emotional and social aspects of life after TL.

SUMMARY:
Total laryngectomy (TL) patients suffer from a myriad of psychological and physiological difficulties following surgery. One of their main difficulties in communication due to problems in speaking. Art therapy offers an alternative means of communication via visual art making and has been shown to reduce psychological distress in cancer patients. Thus the goal of our study is to examine the effect of participating in a group art therapy session on the psychological and physical well being of TL patients. Our design is a quasi-experimental qualitative study with a pre-post design, collecting data with validated questionnaires and self-reports of the participants.

DETAILED DESCRIPTION:
Laryngeal carcinoma (LC) is a cancer that is originated in the larynx which is responsible for three vital functions: the correct passage of air while breathing, closing off the airway during swallowing and voice production. An estimation of around 160,000 new cases of LC are reported worldwide annually, with male predominance. In Israel there are around 200 new cases of LC annually. There are more men than women with the condition and more Arab and Russian immigrants than native Jewish. Laryngeal Cancer can be treated with a combination of surgery, radiotherapy and chemotherapy. The surgical treatment for advanced LC is total laryngectomy (TL). Patients report difficulties adjusting to their stoma, communicating, coughing and eating in public, as well as shame associated with their changed appearance. Many patients state that trying to live the way they did before surgery is frustrating, yet some find hope in striving to get better and "getting back on track". Many patients state they benefited from speaking to other patients about these topics. Psychological well-being is also highly associated with social quality of life.

Laryngectomy patients suffer from dramatic disfigurement. They have a stoma - opening of the trachea at their necks - at a visible location. Patients surveyed at different stages of disease for dissatisfaction with body image and its relation to health related quality of life (HRQOL) reported that they were frequently concerned and dissatisfied with their changed appearance. Dissatisfaction also predicted lesser improvement in HRQOL, recovery and function. Observed disfigurement and dissatisfaction with appearance was shown to be moderated by the sense of social self-efficacy.

A Cochrane review of psychological interventions (C.B.T., dynamic, psycho-education and group interventions) performed with the HNC population showed ambiguous results as to the effects of interventions on improving QOL. This could be due to the difficulty of conducting verbal psychosocial interventions with a population suffering with speech impairments. Art therapy is a means with which patients can express themselves in a non-verbal way, experience creativity, address psychological and social issues, battle addictions and immerse themselves in a feeling of flow. The use of art materials is a sensorial activity that can engage the body in a relatively effortless yet meaningful way.

Studies examining the efficacy of art therapy with cancer patients, demonstrate the decrease of depressive symptoms anxiety and fatigue, moving patient's attention away from worry and pain, improving QOL, and coping capabilities. To the best of our knowledge, there has only been one published study of art therapy with laryngectomy patients. In this article, the art therapist worked with three laryngectomy patients, describing it as an ideal therapy for people with diminished communication capabilities as it provides for a safe arena for them to practice growing communication skills.

Thus, the aim of our study is to examine the psychological changes of post-laryngectomy patients following group art therapy. In order to obtain our study objectives, we propose to conduct a pilot study with Laryngectomy patients at Carmel Medical Center, Haifa, Israel. Our design is a quasi-experimental qualitative study with a pre-post design, collecting data with validated questionnaires and self-reports of the participants.

ELIGIBILITY:
Inclusion Criteria:

* men or women above the age of 18
* TL surgery at least one year ago

Exclusion Criteria:

* Personality disorders that prevent participation in a group.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
The functional assessment of cancer therapy questionnaire (FACT H-N) | 10 minutes
  39 items asking questions about physical, emotional, social and functional well being in the past 7 days

SECONDARY OUTCOMES:
The Center for Epidemiological Studies Depression Scale (CESD R-10) | 5 minutes
  This scale is a self-report measure of depression. The total score is calculated by finding the sum of 10 items. Scores range from 0-40. A score equal to or above 16 indicates a person at risk for clinical depression.

OTHER OUTCOMES:
Art based intervention questionnaire (ABI) | 10 minutes
  41 item questionnaire assessing an individuals experience an art based intervention

REFERENCES:
- [Background] Pereira da Silva A, Feliciano T, Vaz Freitas S, Esteves S, Almeida E Sousa C. Quality of life in patients submitted to total laryngectomy. J Voice. 2015 May;29(3):382-8. doi: 10.1016/j.jvoice.2014.09.002. Epub 2015 Jan 22. PMID 25619472
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] American Society of Clinical Oncology; Pfister DG, Laurie SA, Weinstein GS, Mendenhall WM, Adelstein DJ, Ang KK, Clayman GL, Fisher SG, Forastiere AA, Harrison LB, Lefebvre JL, Leupold N, List MA, O'Malley BO, Patel S, Posner MR, Schwartz MA, Wolf GT. American Society of Clinical Oncology clinical practice guideline for the use of larynx-preservation strategies in the treatment of laryngeal cancer. J Clin Oncol. 2006 Aug 1;24(22):3693-704. doi: 10.1200/JCO.2006.07.4559. Epub 2006 Jul 10. PMID 16832122
- [Background] Dooks P, McQuestion M, Goldstein D, Molassiotis A. Experiences of patients with laryngectomies as they reintegrate into their community. Support Care Cancer. 2012 Mar;20(3):489-98. doi: 10.1007/s00520-011-1101-4. Epub 2011 Feb 6. PMID 21298450
- [Background] Perry A, Casey E, Cotton S. Quality of life after total laryngectomy: functioning, psychological well-being and self-efficacy. Int J Lang Commun Disord. 2015 Jul;50(4):467-75. doi: 10.1111/1460-6984.12148. Epub 2015 Feb 19. PMID 25703153
- [Background] Hagedoorn M, Molleman E. Facial disfigurement in patients with head and neck cancer: the role of social self-efficacy. Health Psychol. 2006 Sep;25(5):643-7. doi: 10.1037/0278-6133.25.5.643. PMID 17014282
- [Background] Semple C, Parahoo K, Norman A, McCaughan E, Humphris G, Mills M. Psychosocial interventions for patients with head and neck cancer. Cochrane Database Syst Rev. 2013 Jul 16;2013(7):CD009441. doi: 10.1002/14651858.CD009441.pub2. PMID 23857592
- [Background] Malchiodi, C. A. (2003). The art and science of art therapy. Handbook of art therapy, 1-5.
- [Background] Nainis N, Paice JA, Ratner J, Wirth JH, Lai J, Shott S. Relieving symptoms in cancer: innovative use of art therapy. J Pain Symptom Manage. 2006 Feb;31(2):162-9. doi: 10.1016/j.jpainsymman.2005.07.006. PMID 16488349
- [Background] Geue K, Goetze H, Buttstaedt M, Kleinert E, Richter D, Singer S. An overview of art therapy interventions for cancer patients and the results of research. Complement Ther Med. 2010 Jun-Aug;18(3-4):160-70. doi: 10.1016/j.ctim.2010.04.001. Epub 2010 May 15. PMID 20688262
- [Background] Anand, S.A. & Anand, V.K. (1997). Art therapy with laryngectomy patients. Art Therapy, 14(2), 109-117.